CLINICAL TRIAL: NCT04983758
Title: Long-term (20-year) Implant Survival and Success Rates in Patients Healthy and Compromised Patients
Brief Title: 20-year Implant Survival in Periodontally Healthy and Compromised Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Turin, Italy (Other)
Responsible Party: Principal Investigator, Mario Roccuzzo, Dr. Mario Roccuzzo, University of Turin, Italy
Other Study IDs: 168/2021
Record Dates: First submitted 2021-07-06; First posted 2021-07-30 (Actual); Last update posted 2021-07-30 (Actual); Status verified 2021-07

CONDITIONS: Dental Implant Failed; Peri-Implantitis; Bone Loss
MeSH Terms: conditions — Peri-Implantitis; Bone Diseases, Metabolic | interventions — Rehabilitation; Dental Implants

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- PHP
  Interventions: Other: Oral Rehabilitation with dental implants
- Moderate PCP
  Interventions: Other: Oral Rehabilitation with dental implants
- Severe PCP
  Interventions: Other: Oral Rehabilitation with dental implants

INTERVENTIONS:
Other: Oral Rehabilitation with dental implants — Patients have been treated with oral dental implants supporting fixed dental prostheses

SUMMARY:
The aim of this study will be to compare the long-term outcomes of sandblasted and acid-etched (SLA) implants in patients previously treated for periodontitis and in periodontally healthy patients (PHP) after a follow-up of at least 20-years.

ELIGIBILITY:
Inclusion Criteria:

* complete edentulism;
* presence of an implant-supported overdenture;
* mucosal diseases;
* alcohol and drug abuse;
* pregnancy;
* uncontrolled metabolic disorders;
* aggressive periodontitis;
* no interest in participating in the study

Exclusion Criteria:

* Everything not as Inclusion Criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients attending the principle investigator (M.R.), a specialist in periodontology, for dental implant therapy between December 1998 and September 2001 were screened for possible inclusion in the study.
Sampling Method: Non-Probability Sample
Enrollment: 149 (Estimated)
Dates: Start 2021-09-01 (Estimated); Primary Completion 2022-09-01 (Estimated); Study Completion 2023-07-01 (Estimated)

PRIMARY OUTCOMES:
Implant survival rate | Baseline; 10-year at the 20-year follow-up examination
  Change in percentage of dental implants in situ / dental implants placed

SECONDARY OUTCOMES:
Marginal Bone loss | Baseline; 10-year at the 20-year follow-up examination
  Changes in mm of the peri-implant marginal bone loss

CONTACTS AND LOCATIONS:
Locations (1):
- University of Torino, Torino, Italy

IPD SHARING:
Plan to Share IPD: No